CLINICAL TRIAL: NCT06182228
Title: The Effectiveness Of Frail Scale And Daily Life Activity Assessments In Determining Postoperative Results In Patients Between 65-85 Years Of Age Which Are Planned For Major Abdominal Surgery
Brief Title: Effectıvenes Of Frail Scale And Daily Lıfe Activity Assesment For Major Abdominal Surgery Patients
Status: Enrolling by invitation | Type: Observational
Sponsor: Uludag University (Other)
Responsible Party: Principal Investigator, Bengü Araz, Principal Investigator, Uludag University
Other Study IDs: 2011-KAEK-26/433
Record Dates: First submitted 2023-11-15; First posted 2023-12-26 (Actual); Last update posted 2024-02-14 (Actual); Status verified 2024-02

CONDITIONS: Frailty
Keywords: Surgical patient
MeSH Terms: conditions — Frailty

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The effectiveness of assessing postoperative outcomes in eldely patients undergoing major abdominal surgery through the Frailty Scale and Katz Activities of Daily Living evaluation is investigated in individuals aged 65-85. The secondary objective is to determine the prevalence of frailty in patients undergoing surgical procedures.

DETAILED DESCRIPTION:
People's life expectancy is increasing rapidly in line with technological progress in the quality of medical care. According to projections by the World Health Organization, it is estimated that by 2030, one in six people worldwide will be aged 60 and above. This figure is expected to reach 2.1 bilion by 2050, with the number of individuals aged 80 and above reaching 426 million.Surgical interventions in elderly patients are associated with increased rates of major complictions, prolonged hospital stays, unplanned readmissions and transfers to rehabilitation center, indicating adverse health outcomes. Therefore, considering the population growth rate, it is inevitable to develop new methods i planning surgical interventions for the elderly. As this point, challenges in surgical planning for individuals fallling under the definition of " frail eldely" become more pronounced. 'Frailty' is a biological syndrome resulting from cumulative declines in multiple physiological systems, leading to vulnerability aganist adverse outcomes, characterized by areduction in reserves and resistance to stress factors. This concept is considered an independent risk factor in predicting and managing postoperative adverse outcomes, beyond aging and comorbidity conditions.Taking into account its determinative impact on surgical outcomes, focusing on the planning of surgical procudures and optimizing postoperative results for patients falling under the definition of "frail elderly" can provide a suitable perspective. Numerous tools have been developed in the literature to measure frailty; however, there is no standardized and approved method for perioperative assessment.The FRAIL Scale, frequently applied in clinical practice to determine levels of frailty, is a practical and straightforward tool. The application, scoring and interpretation of this brief measurement based on interviews are easy. Another easy way to assess the health status of the elderly is to perform a functional assesment that indicates vulnerability and provides objective data. Among the tools used to assess basic activities of daily living, the Katz Index of Independence in Activities of Daily Living is one of the best-known and most commonly used scales clinical practice and research studies.The study aims to determine the effectiveness of FRAIL Scale and Katz Activities of Daily Living assessments in predicting postoperative outcomes, including hospital stay,intensive care needs, readmission rates and duration, reoperation necessity and their associations with morbidity and mortality in patients aged 65-85 undergoing major abdominal surgery and identified in the "frail elderly" stage.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 65-85
* Patients requiring elective major abdominal surgery
* Approval of the informed consent form

Exclusion Criteria:

* Those under the age of 65 and over the age of 85
* Those with cognitive dysfunction
* Those who did not approve of participating in the study
* Patients requiring urgent surgery

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Patients aged 65-85 who underwent major abdominal surgery
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-03-30 (Estimated)

PRIMARY OUTCOMES:
Effectiveness of the FRAIL scale in predicting postoperative outcomes | 1 month
  5 questions of the FRAIL Scale were asked.Questions that evaluated fatigue(How tired have you felt in the last 4 weeks?),resistance(Do you have difficulty climbing 10 flights of stairs on your own, without using any assistive devices, without resting?), wandering (Do you have difficulty walking a few hundred meters on your own and without using an assistive device?), diseases ( How many of the 11 diseases we will list have been told to you by a doctor before as your "disease"? Hypertension, diabetes, cancer (other than minor skin cancer), chronic lung disease, myocardial infarction, congestive heart failure, angina, asthma, arthritis, kidney disease and stroke) and unintentional weight loss (Have you lost 5% of your body weight in the last year?) were given "0" and "1" points. At the end of a total of 5 questions, those who scored 0 points were considered "non-frail", those who scored 1-2 points were considered "pre-frail", and those who scored 3-5 points were considered "frail".

CONTACTS AND LOCATIONS:
Locations (1):
- Uludag Universty, Bursa, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
I have not decided